CLINICAL TRIAL: NCT01663636
Title: SMS Mobile Technology for Vaccine Coverage and Acceptance in Guatemalan Infants
Brief Title: SMS Mobile Technology for Vaccine Coverage and Acceptance
Acronym: Vaxtech
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 12-1144; OPP1061430 (Other)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-06

CONDITIONS: Adherence to Vaccination Schedules
Keywords: vaccines; SMS; mobile phones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SMS Vaccine: Mothers will be sent an SMS message reminding them to come for their scheduled vaccines 1 week prior to the date of 2nd and 3rd doses
  Interventions: Behavioral: SMS message reminding mothers to come for their scheduled vaccines
- Usual care: Mothers under usual care will serve as a control

INTERVENTIONS:
Behavioral: SMS message reminding mothers to come for their scheduled vaccines — Reminder
  Groups: SMS Vaccine

SUMMARY:
To pilot test a mobile phone SMS (Short Message Service) system that will provide periodical messaging texts to mothers or custodians of infants who come for their first dose vaccines within the first 3 months of life to improve timely immunization coverage, vaccine acceptance and ensure vaccine safety monitoring. The intervention will include a "cloud-based" information system alimented by mobile phone data entry at the health post nurse level, that links child vaccination status and is able to remind parents and nurses of the need for next vaccination appointment and provide a system for reporting of adverse events following immunization in the immediate post-vaccination period.

DETAILED DESCRIPTION:
Significance: Vaccine coverage and acceptance in many municipal districts of Guatemala and other low- and middle-income countries are below the acceptable 80% reported at the national level for DPT3 (diphtheria, pertussis, tetanus) and measles vaccines. Despite the considerable effort to introduce new vaccines like Hib (Haemophilus influenzae type B) and rotavirus, in many countries like Guatemala infants do not get immunized on time. Completion of the recommended primary series does not reach beyond 70% of eligible infants by 12 months of age, placing them at risk of disease due to incomplete protection and missing the opportunity to get vaccinated appropriately. Reasons for not getting vaccinated on time include the lack of a system of reminders for the target population, missed opportunities to get vaccinated at the health services due to the lack of vaccine inventories and timely supply of vaccines (including the need for "group sessions for vaccinations" in order to secure the cold chain and vaccine availability).

In addition, monitoring of adverse events following immunization is lacking in most low and middle-income countries. Public acceptance for immunization is based not only on the effectiveness of the vaccine to reduce illness and death, but in the perception of vaccine safety at the population level. To maintain the confidence and acceptance in immunization programs, the reporting and proper response to events following immunization is critical. Allowing parents to notify possible adverse events following immunization provides them with direct access to the health care system to obtain a rapid response for their concerns, but also feedback about the safety of the vaccines and maintain vaccine trust and acceptance. Mobile phone reminders have been used in some populations in high-income countries to recall patients for influenza vaccinations, collect data on asthma dairies, and ensure adherence to antiretroviral therapy. In Guatemala, a country with an estimated population of 14 million inhabitants, there are at least 15 million mobile phones reported in use. At least 4 out of 5 families own and use a mobile phone, and a recent rapid needs assessment from the area of Quetzaltenango showed that at least 48% of mothers from very poor families own and use a mobile phone. The availability of this technology provides with an opportunity to use it as a method to collect information regarding vaccine coverage, use, supply and even monitoring of vaccine safety concerns.

Specific Aims:

1) To pilot test the SMS immunization system that allows immunization reminders to parents and health care workers in order to improve the vaccine timeliness completion rate and overall immunization coverage

Study: 320 infants younger than 3 months of age from municipal districts in Guatemala known to have vaccine coverage rates for DPT3 below 80% and who are coming to the health services for their first dose of vaccine will be recruited for the study. After obtaining consent for participation in the study, the parents will be provided with a mobile phone with SMS capability and instructed on its use. The health care worker will use her mobile device to enter the data on the child including date of birth, mother´s mobile phone number, date of vaccination and vaccines given, and these data will be uploaded into a remote database linked to the mobile phone system.

After the child has been vaccinated the mother or custodian will receive the following SMS notifications:

1. Within 3 days of vaccination an SMS will be send inquiring for any serious or medically relevant adverse events following immunization that the parent will like to report. The response will be uploaded automatically after the parent provides a reply, and will prompt a call from the health care worker if an AEFI (Adverse events following immunization) has been reported into the system.
2. One week before the next scheduled date for 2nd and 3rd dose of vaccines, the parents will automatically receive daily SMS message for 3 consecutive days, instructing them to visit the health care center to vaccinate their children. If the child fails to attend the immunization appointment, the nurse will receive an automatic message one week later reminding her/him to physically recall the child for immunization.

Section II. How will you test it? The intervention will be tested in Guatemala City an area known to have attained vaccine coverage for Pentavalent/DTP3 of only 78% for all its districts in the latest Maternal Infant Health Survey conducted in 2008-2009. The development of the remote data base system as well as the mobile phone base platform will be done in conjunction with local phone companies. Those funds will provide the investment for the development of the software platform, and for the mobile phones and airtime to be given to parents and health care workers.

Essential Data and Outcomes for Phase 1:

1. Rates of completion of primary immunization series in the intervention group including age at completion for 2nd and 3rd doses and rates of missed opportunities for vaccination
2. Satisfaction and feedback about intervention from mother at study completion

ELIGIBILITY:
Inclusion Criteria:

* Infants 1-3 months of age coming for their 1 dose of primary vaccines

Exclusion Criteria:

* Received 1 dose of vaccines, excluding BCG
* No mobile phone with SMS or unable to use SMS at home
* Intent to move from the clinic area in the next 6 months

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants under 12 months of age from Ministry of Health Clinics in Guatemala City
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin J Asturias, MD, Principal Investigator — University of Colorado School of Medicine; Ingrid L Contreras-Roldan, MD, Study Director — University del Valle, Guatemala
Locations (1):
- University del Valle, Guatemala City, Guatemala

REFERENCES:
- [Derived] Domek GJ, Contreras-Roldan IL, O'Leary ST, Bull S, Furniss A, Kempe A, Asturias EJ. SMS text message reminders to improve infant vaccination coverage in Guatemala: A pilot randomized controlled trial. Vaccine. 2016 May 5;34(21):2437-2443. doi: 10.1016/j.vaccine.2016.03.065. Epub 2016 Mar 26. PMID 27026145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents of infants between the ages of 8 and 14 weeks presenting for the first dose of the 3-dose infant primary immunization series were eligible if they owned a mobile phone with SMS text messaging capability and were recruited in 2 pubic health clinics in Guatemala City from April to May of 2013.
Pre-assignment Details: At least one parent had to be literate and able to use SMS technology. Parents were excluded if they were under 18 years of age or if their child had a contraindication to vaccination. Allocation to SMS vaccine (intervention) or usual care (control) was done using a computer generated randomization.
Groups:
- SMS Vaccine: Parent or guardian will be sent an SMS message reminding them to bring in their infant(s) for the infant(s) scheduled vaccines 1 week prior to the date of 2nd and 3rd doses.
- Usual Care: Parent or guardian and their infants who are under usual care (no SMS) will serve as a control group.
Period: Infant SMS Reminder Feasibility Study
Arm/Group | SMS Vaccine | Usual Care
Started | 160 | 161
Completed | 135 | 130
Not Completed | 25 | 31
Not completed — Lost to Follow-up | 25 | 31
Period: Parent SMS Acceptability Assessment
Arm/Group | SMS Vaccine | Usual Care
Started | 135 | 130
Completed | 135 | 130
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Vaccine | Usual Care | Total
Number analyzed (Participants) | 160 | 161 | 321
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 9.7 (1.4) | 9.4 (1.2) | 9.5 (1.3)
Sex/Gender, Customized [Number; unit: participants]
  Male | 76 | 89 | 165
  Female | 84 | 71 | 155
  Missing value | 0 | 1 | 1
Number of Participants who live <16 km from the Clinic [Number; unit: participants]
  Live <16 km from the Clinic | 157 | 160 | 317
  Live =>16 km from the Clinic | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Completion of 3 Doses of Pentavalent Vaccine
Description: Number of children vaccinated with the recommended dose of Pentavalent vaccines according to the age schedule of the National Immunization Program in Guatemala
Time Frame: 8 months of age
Measure: Number; unit: participants
Arm/Group | SMS Vaccine | Usual Care
Number analyzed (Participants) | 160 | 161
participants | 135 | 130

ADVERSE EVENTS:
Time Frame: 1 year
Description: Breaches in confidentiality or inadvertent information releases were monitored.
Arm/Group | SMS Vaccine | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/161
Other Adverse Events (participants affected / at risk) | 0/160 | 0/161

LIMITATIONS AND CAVEATS:
Study was not powered to assess efficacy. SMS texts platform did not have a reporting feature, limiting our ability to confirm message reception. High vaccine visit completion rates made evaluation of an effect challenging.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No